CLINICAL TRIAL: NCT01194817
Title: A Prospective, Randomized Study Comparing Cemented and Cementless Total Knee Replacement: Results of a New Modular Trabecular Metal Tibial Component Using the NexGen System
Brief Title: A Prospective, Randomized Study Comparing Cemented and Cementless Total Knee Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Kevin B. Fricka, MD, Principal Investigator, Anderson Orthopaedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AORI2010-0105
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; total knee replacement; cementless TKA; high flexion; trabecular metal
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented fixation (Other): Nexgen High-Flexion Knee Replacement System using Cemented Fixation
  Interventions: Device: High-Flexion Knee Replacement System using Cemented Fixation
- Cementless fixation (Other): Nexgen High-Flexion Knee Replacement System using Cementless Fixation
  Interventions: Device: High-Flexion Knee Replacement System using Cementless Fixation

INTERVENTIONS:
Device: High-Flexion Knee Replacement System using Cemented Fixation
  Arms: Cemented fixation
Device: High-Flexion Knee Replacement System using Cementless Fixation
  Arms: Cementless fixation

SUMMARY:
The purpose of this study is to compare the the Nexgen knee replacement system using cementless fixation with the same system using cemented fixation. At minimum 2-year follow-up, the hypothesis is that NexGen total knee arthroplasties using cementless and cemented fixation will demonstrate no differences in clinical outcome based on Oxford and Knee Society scores, patient-assessed visual analog pain, clinical complications, radiographic fixation and implant survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of osteoarthritis of the knee
* Patients undergoing primary total knee replacement

Exclusion Criteria:

* Age over 75 years old
* Prior unicondylar knee arthroplasty
* Grossly porotic bone or bone defects requiring bone grafting
* Bone cuts not sufficiently accurate for cementless fixation

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-04; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic analysis | 4 week
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration, and the presence and progression of radiolucent lines between the prosthesis, bone and cement.
Radiographic analysis | 1 year
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration, and the presence and progression of radiolucent lines between the prosthesis, bone and cement.
Radiographic analysis | 2 year
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration, and the presence and progression of radiolucent lines between the prosthesis, bone and cement.
Radiographic analysis | 5 year
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration, and the presence and progression of radiolucent lines between the prosthesis, bone and cement.
Radiographic analysis | 10 year
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration, and the presence and progression of radiolucent lines between the prosthesis, bone and cement.
Radiographic analysis | 15 year
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration, and the presence and progression of radiolucent lines between the prosthesis, bone and cement.
Complications | Date of surgery
  The number and type of adverse events will be monitored to assess safety.
Complications | 4 week
  The number and type of adverse events will be monitored to assess safety.
Complications | 4 month
  The number and type of adverse events will be monitored to assess safety.
Complications | 1 year
  The number and type of adverse events will be monitored to assess safety.
Complications | 2 year
  The number and type of adverse events will be monitored to assess safety.
Complications | 5 year
  The number and type of adverse events will be monitored to assess safety.
Complications | 10 year
  The number and type of adverse events will be monitored to assess safety.
Complications | 15 year
  The number and type of adverse events will be monitored to assess safety.
Radiographic analysis | 4 month
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration, and the presence and progression of radiolucent lines between the prosthesis, bone and cement.

SECONDARY OUTCOMES:
Knee Society Score | 4 week
  A standard clinical evaluation system for reporting results for patients undergoing total knee replacement.
Knee Society Score | 1 year
  A standard clinical evaluation system for reporting results for patients undergoing total knee replacement.
Knee Society Score | 2 year
  A standard clinical evaluation system for reporting results for patients undergoing total knee replacement.
Knee Society Score | 5 year
  A standard clinical evaluation system for reporting results for patients undergoing total knee replacement.
Knee Society Score | 10 year
  A standard clinical evaluation system for reporting results for patients undergoing total knee replacement.
Knee Society Score | 15 year
  A standard clinical evaluation system for reporting results for patients undergoing total knee replacement.
Oxford Knee Score | 4 week
  A patient reported questionnaire for assessing the outcome of knee surgery.
Oxford Knee Score | 1 year
  A patient reported questionnaire for assessing the outcome of knee surgery.
Oxford Knee Score | 2 year
  A patient reported questionnaire for assessing the outcome of knee surgery.
Oxford Knee Score | 5 year
  A patient reported questionnaire for assessing the outcome of knee surgery.
Oxford Knee Score | 10 year
  A patient reported questionnaire for assessing the outcome of knee surgery.
Oxford Knee Score | 15 year
  A patient reported questionnaire for assessing the outcome of knee surgery.
Visual analog pain score | 4 week
  Pain score will be measured from a patient-assessed visual analog pain scale.
Visual analog pain score | 4 month
  Pain score will be measured from a patient-assessed visual analog pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin B Fricka, MD, Principal Investigator — Anderson Orthopaedic Research Institute